CLINICAL TRIAL: NCT04253951
Title: Lung Ultrasound for Early Detection of Silent and Apparent aspiratioN in Infants and Young CHildren With Cerebral Palsy and Other Developmental Disabilities: a New Fast, Safe, Cost-effective Infant-friendly Imaging Tool to Easily Monitor Feeding , Improve Outcomes and Reduce Morbidities (LUNCH)
Brief Title: Lung Ultrasound for Infants' Swallowing Disorders
Acronym: LUNCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Ministry of Health, Italy (Other Government); University of Pisa (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Principal Investigator, Simona Fiori, Principal Investigator, MD, PhD, IRCCS Fondazione Stella Maris
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: LUNCH-2019
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy; Pediatric Neurological Disorder; Developmental Disability
Keywords: abnormal swallowing; infants and young children with neurological impairment; lung ultrasound; apparent aspiration; silent aspiration
MeSH Terms: conditions — Cerebral Palsy; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized parallel-designed controlled trial (Consort checklist, 21), with block randomization (blocks of size 4), in one of 2 groups: 1) LUS-monitored management (LUS-m); 2) Standard care management (SC-m). Both groups will undergo an experimental 6-months follow-up. In the first 3 months, participants will be evaluated a minimum of 1 time per month, in-hospital, for a total of 3 evaluations (T1, T2 and T3), plus baseline (T0).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the clinicians who will perform and score LUS, and the patients' family will be blinded to randomization. The care providers (child neurologist and speech and language pathologist (SLP) will be informed of the result of LUS only in the LUS-m group and will include that result to impact on feeding care (postural, thickening fluids or with drugs available for GERD). LUS results in the SC-m group will be available only at the time of data analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUS-monitored management (LUS-m) (Experimental): In the first 3 months, participants will be evaluated a minimum of 1 time per month, in-hospital, for a total of 3 evaluations (T1, T2 and T3), plus baseline (T0). At any time point, they will undergo at least one LUS-monitored (before and after) feeding trial (different consistencies might be tested in separate repeated trials according to clinical evaluation). A further LUS evaluation will be performed at a distance of 3 hours, before the next meal to check for resolution of after-meal abnormalities.
  Interventions: Diagnostic Test: Lung Ultrasound (LUS)-monitored feeding trial
- Standard care management (SC-m) (Sham Comparator): Sham protocol with LUS performed at the same timepoints. LUS results in the SC-m group will be available only at the time of data analyses for comparison by investigators. They will not be used for clinical decisions.
  Interventions: Diagnostic Test: Lung Ultrasound (LUS)-monitored feeding trial

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound (LUS)-monitored feeding trial — LUS-monitored (before and after) feeding trial (different consistencies might be tested in separate repeated trials according to clinical evaluation). A further LUS evaluation will be performed at a distance of 3 hours, before the next meal to check for resolution of after-meal abnormalities. All pulmonary fields will be explored according to semeiotics and previous literature.

SUMMARY:
The aim is to test the effectiveness of lung ultrasound (LUS) in the dynamic assessment of aspiration related to abnormal swallowing in infants and young children with neurological impairment (cerebral palsy/developmental disabilities). Neither standardized measure is available, nor protocols for invasive fibre-optic endoscopic examination of swallowing (FEES) and x-Ray videofluoroscopic swallowing study (VFSS) to be used in such population. LUS offers several advantages: time saving for aspiration diagnosis; safeness (neither invasiveness nor radiation); repeatability with different meal consistencies or to monitor interventions efficacy; cost-effectiveness; savings of x-Ray exposition (compared to VFSS). All these advantages may lead infants to improve clinical behavioural and neurological outcomes and reduce stressful interactions with caregivers, and to reduce morbidities and hospitalization costs for respiratory and non-respiratory complications related to swallowing disorders.

DETAILED DESCRIPTION:
The dynamic use of LUS for monitoring feeding related aspiration can be effective in detecting meal-related pulmonary abnormalities in neurologically impaired infants and that LUS-management will improve medical/neurological/behavioural status, and reduce chronic pain/discomfort and stress for caregivers. LUS effectiveness is expected to reduce the need for x-Ray, invasive and more expensive techniques (VFSS and FEES). Results may be translated into clinical practice in the management of swallowing disorders in a very vulnerable population, by reducing invasiveness, possible x-Ray early exposition risks, costs, medical complications, and by assessing risk categories based on neuroimaging MRI markers, to rationalize prevention and intervention.

Preliminary data. LUS examinations have been performed on 6 infants with neurological impairment (mean age 15 ± 8 months; Gross Motor Function Classification System (GMFCS) range 2-5, median=4) and in 3 healthy infants (mean age 25 ± 3 months) before and right after a meal. A LUS score ranging from 0 to 18 was established, according to previous literature (0= normal pattern, 1= separated B-lines, 2= confluent B-lines or B-lines with pleural alterations, 3= consolidations; the score 0-3 was then calculated in all 6 thoracic scanning areas and summed up). In the 6 infants with neurological impairment, at paired sample t test, LUS score changed before and after meal (pre-meal 2.50±2.95 vs post-meal 5.17±3.25, p=0.01), with very large effect size (Cohen d=1.6). No change was detected in the control group. Changes in LUS score pre and post-meal correlated with GMFCS (p=0.03, r=0.64) and with adapted Eating and Drinking Ability Classification System (EDACS) scores (p=0.04, r=0.59), as more severe clinical pictures resulted in worse LUS scores. The LUS score pre- meal was worse in infants with neurological impairment compared to controls (2.50±2.95 vs 0.67±0.58, p=0.14). Results make LUS extremely promising as a tool to monitor pulmonary aeration changes in infants with neurological impairment. Feasibility of dorsal and ventral oromotor tract reconstruction has been tested in an infant with neurological impairment.

Specific Aim 1:

* To establish the feasibility and effectiveness of LUS-guided management in the detection of aspiration related to swallowing disorders in children with cerebral palsy and other developmental disabilities, determining advantages of LUS-guided management over standard care on medical (respiratory illness and growth rate) LUS findings themselves and behavioural/neurological outcomes
* To compare diagnostic accuracy of LUS versus X-ray VFSS and invasive FEES

Specific Aim 2:

- To determine specific parameters to estimate aspiration entity by LUS (eg cut-off values for the diagnosis of clinically significant silent or overt aspiration, responsiveness of LUS monitoring to medical, postural or food consistencies adaptation) and their relationship with standardised clinical feeding evaluation and medical/behavioural/neurological measures in order to define risk groups for aspiration

Specific Aim 3:

* To evaluate other applications/potentialities of LUS in children with cerebral palsy and other developmental disabilities.
* To uncover the impact of brain abnormalities detected by brain MRI on LUS findings, for establishing risk categories for unsafe swallowing disorders on early imaging markers, and potential clinical recommendations for early management.

Experimental Design Aim 1:

Double-blinded randomized parallel-designed controlled trial (Consort checklist), with block randomization (blocks of size 4), in one of 2 groups: 1) LUS-monitored management (LUS-m); 2) Standard care management (SC-m). Both groups will undergo an experimental 6-months follow-up. In the first 3 months, participants will be evaluated a minimum of 1 time per month, in-hospital, for a total of 3 evaluations (T1, T2 and T3), plus baseline (T0). At any time point, they will undergo at least one LUS-monitored (before and after) feeding trial (different consistencies might be tested in separate repeated trials according to clinical evaluation). A further LUS evaluation will be performed at a distance of 3 hours, before the next meal to check for resolution of after-meal abnormalities. Both the clinicians who will perform and score LUS, and the patients' family will be blinded to randomization. The child neurologist and the speech and language pathologist (SLP) will be informed of the result of LUS only in the LUS-m group and will include that result to impact on feeding care (postural, thickening fluids or with drugs available for GERD). LUS results in the SC-m group will be available only at the time of data analyses. All meals will be monitored by pulse-oximetry and video recording. A further 6-months LUS-monitored and clinical assessment (T4) will be delivered for collecting outcome measures in both treatment groups. At T0, T3 and T4 time points, infants will perform standardized medical/behavioural/neurological, chronic pain/discomfort assessments. At T0 and T4, a blood sample will be collected, to evaluate general and nutritional status, and a quantitative ultrasound (QUS) will be performed to evaluate bone density. A parent stress questionnaire (Parenting Stress Index (PSI)) will be delivered (T0, T3 and T4). Between T0 and T4, parents will be asked to fill a respiratory infection-diary for respiratory illness rate calculation. VFSS and FEES data will be collected, compared in frequency of execution between groups, and their results will be compared to LUS findings. Primary and secondary outcome measures will be collected at both T3 (short-term) and T4 (long-term).

Experimental Design Aim 2:

Aim 2 is based on the same design as Aim 1. We will explore the frequency, severity and distribution of basal and feeding related LUS parameters and their relationship with clinical (feeding assessment/medical/behavioural/neurological/chronic pain) measures, interventions (postural, thickening fluids or with drugs available for GERD), inter- and intra- group at any time point.

Other possible applications of LUS in the enrolled population will be collected (e.g. pneumonia detection and monitoring).

Experimental Design Aim 3:

Brain MRI is a clinical procedure in the diagnostic approach to children with neurological impairment. Brain abnormalities and corticobulbar tract integrity for lips, tongue, larynx motor and sensory control will be checked to uncover the neural circuits that may underlay swallowing problems leading to silent or overt aspiration and pulmonary risk estimated by LUS. Brain lesions topography and severity will be assessed by using a standardized MRI acquisition protocol according to the diagnostic procedure in use at Stella Maris Scientific Institute MRI Lab. Diffusion-weighted Imaging (DWI) will be used with the aim of revealing structural integrity and connectivity along white matter tracts involved in swallowing.

Expected outcomes:

the LUS-m group having better outcomes, at short- and long-term, including: having lower rate of pulmonary illness, better growth curve, reduction of execution rate of VFSS/FEES. Also, better results at blood sample and bone metabolism, lower pain indices, better scores at neurological/behavioural clinical measures, and less stressful interaction with caregivers.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy or abnormal muscular tone at any age between 0-3 years of life due disorders other than cerebral palsy;
* motor developmental delay assessed by a quantitative scale for infants and young children development (<5 sd according to age)
* in absence of the previous clinical indices, if there is the clinical suspicion of GERD or dysphagia based on clinical symptoms
* a brain MRI acquisition done before or programmed prior the end of the study period as part of their diagnostic procedure.

Exclusion Criteria:

* epileptic spasm
* drugs for muscle tone abnormalities or GERD introduced or modified less than 3 weeks before potential enrollment

Ages: 3 Weeks to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
respiratory | long term (T4, at 6 months)
  respiratory illness rate (including pneumonia, wheezing, chronic cough, and apnoea rate)
respiratory | short term (T3, at 3 months)
  respiratory illness rate (including pneumonia, wheezing, chronic cough, and apnoea rate)
growth | long term (T4, at 6 months)
  growth rate
growth | short term (T3, at 3 months)
  growth rate
invasive diagnostic | long term (T4, at 6 months)
  VFSS/FEES execution rates
invasive diagnostic | short term (T3, at 3 months)
  VFSS/FEES execution rates

SECONDARY OUTCOMES:
change from baseline laboratory exam at 6 months | baseline-long term (T4, at 6 months)
  blood cells count
change from baseline laboratory exam at 6 months | baseline-long term (T4, at 6 months)
  reticulocytes count
change from baseline laboratory exam at 6 months | baseline- long term (T4, at 6 months)
  total serum protein
change from baseline laboratory exam at 6 months | baseline- long term (T4, at 6 months)
  ferritin
chronic pain assessment | short term (T3, at 3 months)
  parents-report measure (Non-communicating Children's Pain Checklist, NCCPC), with scores ranging from 0 to 90, with higher scores corresponding to worse outcome
chronic pain assessment | long term (T4, at 6 months)
  parents-report measure (Non-communicating Children's Pain Checklist, NCCPC), with scores ranging from 0 to 90, with higher scores corresponding to worse outcome
parents' stress | long term (T4, at 6 months)
  Parenting Stress Index questionnaire (PSI), with scores ranging from 0 to 120 including 4 domains, with higher scores corresponding to worse outcome

OTHER OUTCOMES:
neurological outcome | short term (T3, at 3 months) and long term (T4, at 6 months)
  Hammersmith Infant Neurological Examination (HINE), with scores ranging from 0 to 78, with higher scores corresponding to better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simona Fiori, MD, PhD, Principal Investigator — IRCCS Fondazione Stella Maris
Locations (2):
- Italy (2):
  - IRCCS Fondazione Stella Maris, Tirrenia, Tuscany
  - IRCCS Fondazione Stella Maris, Pisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Srivastava R, Jackson WD, Barnhart DC. Dysphagia and gastroesophageal reflux disease: dilemmas in diagnosis and management in children with neurological impairment. Pediatr Ann. 2010 Apr;39(4):225-31. doi: 10.3928/00904481-20100318-07. No abstract available. PMID 20411900
- [Result] Fitzgerald DA, Follett J, Van Asperen PP. Assessing and managing lung disease and sleep disordered breathing in children with cerebral palsy. Paediatr Respir Rev. 2009 Mar;10(1):18-24. doi: 10.1016/j.prrv.2008.10.003. Epub 2009 Jan 23. PMID 19203740
- [Result] Arvedson J, Rogers B, Buck G, Smart P, Msall M. Silent aspiration prominent in children with dysphagia. Int J Pediatr Otorhinolaryngol. 1994 Jan;28(2-3):173-81. doi: 10.1016/0165-5876(94)90009-4. PMID 8157416
- [Result] Blackmore AM, Bear N, Blair E, Gibson N, Jalla C, Langdon K, Moshovis L, Steer K, Wilson AC. Factors Associated with Respiratory Illness in Children and Young Adults with Cerebral Palsy. J Pediatr. 2016 Jan;168:151-157.e1. doi: 10.1016/j.jpeds.2015.09.064. Epub 2015 Oct 29. PMID 26520916
- [Result] Pillai Riddell RR, Stevens BJ, McKeever P, Gibbins S, Asztalos L, Katz J, Ahola S, Din L. Chronic pain in hospitalized infants: health professionals' perspectives. J Pain. 2009 Dec;10(12):1217-25. doi: 10.1016/j.jpain.2009.04.013. Epub 2009 Jun 21. PMID 19541547
- [Result] Benfer KA, Weir KA, Boyd RN. Clinimetrics of measures of oropharyngeal dysphagia for preschool children with cerebral palsy and neurodevelopmental disabilities: a systematic review. Dev Med Child Neurol. 2012 Sep;54(9):784-95. doi: 10.1111/j.1469-8749.2012.04302.x. Epub 2012 May 14. PMID 22582745
- [Result] van den Engel-Hoek L, Erasmus CE, van Hulst KC, Arvedson JC, de Groot IJ, de Swart BJ. Children with central and peripheral neurologic disorders have distinguishable patterns of dysphagia on videofluoroscopic swallow study. J Child Neurol. 2014 May;29(5):646-53. doi: 10.1177/0883073813501871. Epub 2013 Sep 9. PMID 24022110
- [Result] Calvo I, Conway A, Henriques F, Walshe M. Diagnostic accuracy of the clinical feeding evaluation in detecting aspiration in children: a systematic review. Dev Med Child Neurol. 2016 Jun;58(6):541-53. doi: 10.1111/dmcn.13058. Epub 2016 Feb 9. PMID 26862075
- [Result] Cichero J, Nicholson T, Dodrill P. Liquid barium is not representative of infant formula: characterisation of rheological and material properties. Dysphagia. 2011 Sep;26(3):264-71. doi: 10.1007/s00455-010-9303-3. Epub 2010 Sep 10. PMID 20830598
- [Result] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518
- [Result] Uhm KE, Yi SH, Chang HJ, Cheon HJ, Kwon JY. Videofluoroscopic swallowing study findings in full-term and preterm infants with Dysphagia. Ann Rehabil Med. 2013 Apr;37(2):175-82. doi: 10.5535/arm.2013.37.2.175. Epub 2013 Apr 30. PMID 23705111
- [Result] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Result] Raimondi F, Migliaro F, Sodano A, Umbaldo A, Romano A, Vallone G, Capasso L. Can neonatal lung ultrasound monitor fluid clearance and predict the need of respiratory support? Crit Care. 2012 Nov 14;16(6):R220. doi: 10.1186/cc11865. PMID 23151314
- [Result] Raimondi F, Migliaro F, Sodano A, Ferrara T, Lama S, Vallone G, Capasso L. Use of neonatal chest ultrasound to predict noninvasive ventilation failure. Pediatrics. 2014 Oct;134(4):e1089-94. doi: 10.1542/peds.2013-3924. Epub 2014 Sep 1. PMID 25180278
- [Result] Gargani L, Volpicelli G. How I do it: lung ultrasound. Cardiovasc Ultrasound. 2014 Jul 4;12:25. doi: 10.1186/1476-7120-12-25. PMID 24993976
- [Result] Balk DS, Lee C, Schafer J, Welwarth J, Hardin J, Novack V, Yarza S, Hoffmann B. Lung ultrasound compared to chest X-ray for diagnosis of pediatric pneumonia: A meta-analysis. Pediatr Pulmonol. 2018 Aug;53(8):1130-1139. doi: 10.1002/ppul.24020. Epub 2018 Apr 26. PMID 29696826
- [Result] Brenner D, Elliston C, Hall E, Berdon W. Estimated risks of radiation-induced fatal cancer from pediatric CT. AJR Am J Roentgenol. 2001 Feb;176(2):289-96. doi: 10.2214/ajr.176.2.1760289. PMID 11159059
- [Result] Goh YR, Choi JY, Kim SA, Park J, Park ES. Comparisons of severity classification systems for oropharyngeal dysfunction in children with cerebral palsy: Relations with other functional profiles. Res Dev Disabil. 2018 Jan;72:248-256. doi: 10.1016/j.ridd.2017.12.002. Epub 2017 Dec 7. PMID 29223113
- [Result] Pandis N, Chung B, Scherer RW, Elbourne D, Altman DG. CONSORT 2010 statement: extension checklist for reporting within person randomised trials. BMJ. 2017 Jun 30;357:j2835. doi: 10.1136/bmj.j2835. PMID 28667088
- [Result] Liegeois FJ, Butler J, Morgan AT, Clayden JD, Clark CA. Anatomy and lateralization of the human corticobulbar tracts: an fMRI-guided tractography study. Brain Struct Funct. 2016 Jul;221(6):3337-45. doi: 10.1007/s00429-015-1104-x. Epub 2015 Sep 28. PMID 26411871
- [Result] Erasmus CE, van Hulst K, Rotteveel JJ, Willemsen MA, Jongerius PH. Clinical practice: swallowing problems in cerebral palsy. Eur J Pediatr. 2012 Mar;171(3):409-14. doi: 10.1007/s00431-011-1570-y. Epub 2011 Sep 20. PMID 21932013
- [Result] O'Rourke D. The measurement of pain in infants, children, and adolescents: from policy to practice. Phys Ther. 2004 Jun;84(6):560-70. No abstract available. PMID 15161421
- [Result] Bouhemad B, Mongodi S, Via G, Rouquette I. Ultrasound for "lung monitoring" of ventilated patients. Anesthesiology. 2015 Feb;122(2):437-47. doi: 10.1097/ALN.0000000000000558. No abstract available. PMID 25501898
- [Derived] Fiori S, Scaramuzzo RT, Moretti E, Amador C, Controzzi T, Martinelli A, Filippi L, Guzzetta A, Gargagni L. LUNCH-Lung Ultrasound for early detection of silent and apparent aspiratioN in infants and young CHildren with cerebral palsy and other developmental disabilities: study protocol of a randomized controlled trial. BMC Pediatr. 2022 Jun 23;22(1):360. doi: 10.1186/s12887-022-03413-z. PMID 35739502